CLINICAL TRIAL: NCT02501473
Title: Phase 1/2 Study of Intratumoral G100 With Or Without Pembrolizumab or Rituximab In Patients With Follicular Non-Hodgkin's Lymphoma
Brief Title: Study of Intratumoral G100 With Or Without Pembrolizumab or Rituximab In Participants With Follicular Non-Hodgkin's Lymphoma (MK-3475-174/IMDZ-G142)
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Business reasons
Sponsor: Immune Design, a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3475-174; IMDZ-G142 (Other: Immune Design Protocol Number); MK-3475-174 (Other: Merck Protocol Number); 2015-005382-23 (EudraCT Number)
Record Dates: First submitted 2015-07-08; First posted 2015-07-17 (Estimated); Results first posted 2020-09-09 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2020-08

CONDITIONS: Follicular Low Grade Non-Hodgkin's Lymphoma
Keywords: follicular lymphoma; FL; low-grade lymphoma; Non-Hodgkin's Lymphoma; follicular NHL; Marginal Zone
MeSH Terms: conditions — Lymphoma, Follicular; Lymphoma, Non-Hodgkin | interventions — TLR4 agonist G100; pembrolizumab; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Part 1: Local Radiation + G100 5μg/tumor (Experimental): Part 1: Local radiation and G100 [glucopyranosyl lipid A stable emulsion, GLA-SE] at 5μg/tumor administered intratumorally (IT) into accessible tumors for up to 8 weeks.
  Interventions: Drug: G100
- Part 1: Local Radiation + G100 10μg/tumor (Experimental): Part 1: Local radiation and G100 at 10μg/tumor administered IT into accessible tumors for up to 8 weeks.
  Interventions: Drug: G100
- Part 2: Local Radiation + G100 10μg/tumor (Experimental): Part 2: Local radiation and G100 at 10μg/tumor administered IT into accessible tumors for up to 8 weeks.
  Interventions: Drug: G100
- Part 2: Local Radiation + G100 10μg/tumor+Pembrolizumab 200mg (Experimental): Part 2: Local radiation and G100 at 10μg/tumor administered IT into accessible tumors for up to 8 weeks; pembrolizumab 200mg intravenously (IV) administered every 3 weeks (Q3W) IV for up to 2 years.
  Interventions: Drug: G100; Drug: Pembrolizumab
- Part 2: Local Radiation, G100 20 μg/tumor in Large Tumors (Experimental): Part 2: Local radiation and G100 at 20 μg/tumor administered IT into accessible large tumors [injectable lymphoma mass(es) ≥ 4 cm in total size] for up to 8 weeks.
  Interventions: Drug: G100
- Part 3: Local Radiation + G100 20μg/tumor (Experimental): Part 3: Local radiation and G100 at 20μg/tumor administered IT into accessible tumors for up to 8 weeks.
  Interventions: Drug: G100
- Part 4: G100 20μg/tumor and pembrolizumab 200mg (Experimental): Part 4: G100 at 20μg/tumor administered IT into accessible tumors for up to 8 weeks and pembrolizumab 200mg IV and administered Q3W for up to 2 years.
  Interventions: Drug: G100; Drug: Pembrolizumab
- Part 5: G100 + Rituximab 375mg/m^2 (Experimental): Part 5: G100 at 20, 40, 60, or 80μg/tumor administered IT for up to 6 weeks and rituximab administered as an IV infusion at 375mg/m^2 on Day 0 and then QW for up to 3 weeks.
  Interventions: Drug: G100; Drug: Rituximab

INTERVENTIONS:
Drug: G100 — GLA is a fully synthetic toll-like receptor-4 (TLR4) agonist
  Other Names: glucopyranosyl lipid A stable emulsion, GLA-SE
Drug: Pembrolizumab — PD-1 Inhibitor
  Other Names: Keytruda; MK-3475
  Arms: Part 2: Local Radiation + G100 10μg/tumor+Pembrolizumab 200mg; Part 4: G100 20μg/tumor and pembrolizumab 200mg
Drug: Rituximab — Rituximab (anti-CD20 antibody)
  Arms: Part 5: G100 + Rituximab 375mg/m^2

SUMMARY:
This is a Phase 1/2 open label trial of G100 in participants with low grade Non-Hodgkin's Lymphoma (NHL). G100 is composed of glucopranosyl lipid A in a stable emulsion and is a potent TLR4 (toll-like receptor-4) agonist. G100 will be administered by direct injection (intratumorally) into tumors of low grade NHL with or without standard low dose radiation therapy. Preclinical models and clinical studies in other cancers such as Merkel cell carcinoma have demonstrated that G100 administered in this manner can alter the tumor microenvironment, activate dendritic cells, T cells and other immune cells and induce systemic anti-tumor immune responses. In this trial, the safety, immunogenicity, and preliminary clinical efficacy of G100 will be examined alone or with pembrolizumab.

DETAILED DESCRIPTION:
This is a multi-center Phase 1/2 open label trial of intratumoral G100 in participants with low grade NHL. Eligible participants with NHL will be enrolled and receive G100 to an accessible tumor mass. Clinical response will be evaluated in the injected tumor and systemic (abscopal) responses will be evaluated in distal areas involved with tumor.

The study will be conducted in 5 parts. In Part 1, Dose Escalation, 2 sequentially enrolled cohorts of participants will be treated at one of 2 dose levels of G100 using a standard escalation design. In this portion of the study, both follicular and marginal zone NHL will be eligible. In Part 2, 2 groups of participants with follicular NHL may be examined. One group will be randomly assigned to receive either single agent G100 intratumorally at the maximum safe dose determined in Part 1 following local radiation or will receive the same treatment regimen sequentially administered with pembrolizumab. A second treatment group may be explored if the safety profile in Part 1 is acceptable. In this optional group, participants with injectable tumors of 4 cm or greater would be enrolled and treated with a higher dose of G100. In Part 3, expansion of a higher dose (20µg of G100) in participants with follicular NHL will be enrolled to receive local radiation therapy and intratumoral G100. In Part 4, Dose Escalation and Expansion, a dose of 20µg of G100 will be examined as a treatment of 1 or more tumors (up to 4) with pembrolizumab in order to establish safety and examine clinical and biomarker responses in participants receiving increasing total systemic doses of G100 and Part 5, will evaluate standard induction therapy with rituximab (anti-CD20) in combination of escalating doses of intratumoral G100 in single tumors.

The primary goal of this study is to determine the safety and tolerability of different doses of G100 when administered by intratumoral injection. The development of anti-tumor immune responses and preliminary evidence of clinical responses in local and distal tumor sites will also be examined.

ELIGIBILITY:
Inclusion Criteria:

1. Follicular low-grade NHL:

   * In Part 1-3: either treatment naïve (except for France) OR relapsed or refractory following at least one prior treatment.
   * In Part 4, enrollment is limited to relapsed OR refractory follicular NHL participants.
   * In Part 5, enrollment will include relapsed and refractory CD20+ follicular NHL following at least one but not more than 2 prior treatments.
2. Tumor mass(es) accessible for intratumoral injection

   * For Part 1-3, are being considered for local radiation therapy and at least one additional site of disease outside the radiation field for assessment of distal (abscopal) response.
   * For Part 4 and 5, radiation therapy is omitted. Measurable tumor mass(es) accessible for intratumoral injection must be present for treatment and assessment of response.
3. ≥ 18 years of age
4. Life expectancy of ≥ 6 months per the investigator
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
6. Electrocardiogram (ECG) without evidence of clinically significant arrhythmia or ischemia
7. If female of childbearing potential (FCBP), willing to undergo pregnancy testing and agrees to use two methods of birth control or is considered highly unlikely to conceive during the dosing period and for three months after last study treatment, or if receiving pembrolizumab, four months after last treatment
8. If male and sexually active with a FCBP, must agree to use highly effective contraception such as latex condom or is sterile (e.g. following a surgical procedure) during the dosing period and for three months after last study treatment, or if receiving pembrolizumab, four months after last treatment

Exclusion Criteria:

1. Cancer therapies, including chemotherapy, radiation (non-study regimen related), biologics or kinase inhibitors, granulocyte-colony stimulating factor (G-CSF) or granulocyte/monocyte-colony stimulating factor (GM-CSF) within 4 weeks prior to the first scheduled G100 dose
2. Investigational therapy within 4 weeks prior to G100 dosing
3. Prior administration of other intratumoral immunotherapeutics
4. Inadequate organ function including:

   1. Marrow: Peripheral blood leukocyte count (WBC) < 3000/mm^3, absolute neutrophil count ≤ 1500/mm^3, platelets < 75000/mm^3, or hemoglobin < 10 gm/dL
   2. Hepatic: alanine aminotransferase (ALT), and aspartate aminotransferase (AST) > 2.5 x Upper Limit of Normal (ULN), total serum bilirubin > 1.5 x ULN (participants with Gilbert's Disease may be included if their total bilirubin is ≤3.0 mg/dL)
   3. Renal: Creatinine > 1.5x ULN
   4. Other: INR (international normalized ratio) or partial thromboplastin time (PTT) >1.5 x ULN
5. Significant immunosuppression from:

   1. Concurrent, recent (≤ 4 weeks ago) or anticipated treatment with systemic corticosteroids at any dose, or
   2. Other immunosuppressive medications such as methotrexate, cyclosporine, azathioprine or conditions such as common variable hypogammaglobulinemia
6. Pregnant or nursing
7. Myocardial infarction within 6 months of study initiation, active cardiac ischemia or New York Heart Association (NYHA) Grade III or IV heart failure
8. History of other cancer within 2 years (except non-melanoma cutaneous malignancies and cervical carcinoma in situ)
9. Recent (<1 week ago) clinically significant infection, active tuberculosis or evidence of active hepatitis B, hepatitis C or HIV infection
10. Central nervous system involvement with lymphoma, including parenchymal and leptomeningeal disease.
11. Significant autoimmune disease, including active non-infectious pneumonitis, with the exception of alopecia, vitiligo, hypothyroidism or other conditions that have never been clinically active or were transient and have completely resolved and require no ongoing therapy
12. Psychiatric, other medical illness or other condition that in the opinion of the principal investigator (PI) prevents compliance with study procedures or ability to provide valid informed consent
13. History of significant adverse or allergic reaction to any component of G100 and, if enrolled in Part 2 or Part 4, pembrolizumab and/or any of its excipients, and if enrolled in Part 5, anti-CD20 antibodies including rituximab and/or any of its excipients
14. Use of anti-coagulant agents or history a significant bleeding diathesis. (If a superficial lymph node or subcutaneous mass is to be injected, participants on agents such as non-steroidal anti-inflammatory drugs (NSAIDs), aspirin, or clopidogrel are eligible and these agents do not have to be withheld. For procedures with moderate or significant risk of bleeding, long-acting agents such as aspirin or clopidogrel should be discussed with the Medical Monitor and may need to be discontinued before G100 therapy.

    For participants enrolled in Part 2 or Part 4 with the potential to receive pembrolizumab:
15. History of (non-infectious) pneumonitis that required steroids or has current pneumonitis or interstitial lung disease
16. Received a live virus vaccine within 30 days of planned study start
17. Has undergone prior allogeneic hematopoietic stem cell transplantation within the last 5 years. (Participants who have had a transplant greater than 5 years ago are eligible as long as there are no symptoms of graft vs. host disease [GVHD]).
18. Has had an allogeneic tissue/solid organ transplant
19. Has received prior therapy with an anti-PD-1, anti-programmed death ligand (PD-L)1, or anti-PD-L2 agent or if the participant has previously participated in Merck MK-3475 clinical trials or was previously treated with an agent directed to another stimulatory or co-inhibitory T-cell receptor (e.g., CTLA-4, OX 40, CD137) and was discontinued from that treatment due to a Grade 3 or higher immune-related adverse event.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2016-02-03 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2019-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Knapp, Study Director — Clinical Trial Manager

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Halwani AS, Panizo C, Isufi I, Herrera AF, Okada CY, Cull EH, Kis B, Chaves JM, Bartlett NL, Ai W, de la Cruz-Merino L, Bryan LJ, Houot R, Linton K, Briones J, Chau I, von Keudell GR, Lu H, Yakovich A, Chen M, Meulen Jh T, Yurasov S, Hsu FJ, Flowers CR. Phase 1/2 study of intratumoral G100 (TLR4 agonist) with or without pembrolizumab in follicular lymphoma. Leuk Lymphoma. 2022 Apr;63(4):821-833. doi: 10.1080/10428194.2021.2010057. Epub 2021 Dec 6. PMID 34865586

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled in the study at clinical sites in the United States and Europe.
Pre-assignment Details: Part 5, G100 plus Rituximab, Dose Escalation: 12 to 24 participants were planned; no participant was enrolled or dosed.
Groups:
- Part 2: Local Radiation, G100 20 μg/Tumor in Large Tumors: Part 2: Local radiation and G100 at 20 μg/tumor administered IT into accessible large tumors (injectable lymphoma mass(es) ≥ 4 cm in total size) for up to 8 weeks.
- Part 5: G100 + Rituximab 375 mg/m^2: Part 5: G100 administered at 20, 40, 60, or 80 μg/tumor for up to 6 weeks and rituximab (anti-CD20 antibody). Rituximab dose administered as an IV infusion at 375 mg/m^2 administered on Day 0 and then once weekly for 4 doses up to 3 weeks.
Period: Overall Study
Arm/Group | Part 1: Local Radiation + G100 5μg/Tumor | Part 1: Local Radiation + G100 10μg/Tumor | Part 2: Local Radiation + G100 10μg/Tumor | Part 2: Local Radiation + G100 10μg/Tumor+Pembrolizumab 200mg | Part 2: Local Radiation, G100 20 μg/Tumor in Large Tumors | Part 3: Local Radiation + G100 20μg/Tumor | Part 4: G100 20μg/Tumor and Pembrolizumab 200mg | Part 5: G100 + Rituximab 375 mg/m^2
Started | 3 | 3 | 13 | 14 | 4 | 14 | 1 | 0
Treated | 3 | 3 | 13 | 13 | 4 | 14 | 1 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 3 | 3 | 13 | 14 | 4 | 14 | 1 | 0
Not completed — Study Terminated | 2 | 3 | 7 | 9 | 2 | 10 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 3 | 3 | 2 | 2 | 0 | 0
Not completed — Death | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Not completed — Reason not specified | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The analysis population included all randomized and treated participants. Part 5, G100 plus Rituximab, Dose Escalation: 12 to 24 participants were planned; no participant was enrolled or dosed.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1: Local Radiation + G100 5μg/Tumor | Part 1: Local Radiation + G100 10μg/Tumor | Part 2: Local Radiation + G100 10μg/Tumor | Part 2: Local Radiation + G100 10μg/Tumor+Pembrolizumab 200mg | Part 2: Local Radiation, G100 20 μg/Tumor in Large Tumors | Part 3: Local Radiation + G100 20μg/Tumor | Part 4: G100 20μg/Tumor and Pembrolizumab 200mg | Total
Number analyzed (Participants) | 3 | 3 | 13 | 13 | 4 | 14 | 1 | 51
Age, Continuous [Mean (Standard Deviation); unit: Years] | 54.0 (13.45) | 56.3 (16.07) | 60.2 (10.26) | 57.6 (10.98) | 59.3 (5.85) | 63.9 (8.74) | NA (NA) — Age not reported due to risk of identification of a person. | 60.3 (10.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3 | 3 | 1 | 5 | 1 | 16
  Male | 2 | 1 | 10 | 10 | 3 | 9 | 0 | 35
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1 | 3 | 0 | 0 | 0 | 5
  Not Hispanic or Latino | 2 | 2 | 12 | 10 | 4 | 13 | 1 | 44
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 2
  White | 2 | 3 | 11 | 12 | 2 | 12 | 1 | 43
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1 | 1 | 1 | 1 | 0 | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With an Adverse Event (AE)
Description: An adverse event (AE) is defined as any unfavorable and unintended sign including an abnormal laboratory finding, symptom or disease associated with the use of a medical treatment or procedure, regardless of whether it is considered related to the medical treatment or procedure, that occurs during the course of the study.
Time Frame: Up to approximately 42 months
Population: The analysis population included all enrolled participants who received at least 1 injection of G100 after standard local radiation.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Local Radiation + G100 5μg/Tumor | Part 1: Local Radiation + G100 10μg/Tumor | Part 2: Local Radiation + G100 10μg/Tumor | Part 2: Local Radiation + G100 10μg/Tumor+Pembrolizumab 200mg | Part 2: Local Radiation, G100 20 μg/Tumor in Large Tumors | Part 3: Local Radiation + G100 20μg/Tumor | Part 4: G100 20μg/Tumor and Pembrolizumab 200mg
Number analyzed (Participants) | 3 | 3 | 13 | 13 | 4 | 14 | 1
Participants | 3 | 3 | 13 | 13 | 4 | 14 | 1

2. Primary Outcome: Number of Participants Who Discontinued Study Drug Due to an Adverse Event
Description: as for outcome 1
Time Frame: Up to approximately 105 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Local Radiation + G100 5μg/Tumor | Part 1: Local Radiation + G100 10μg/Tumor | Part 2: Local Radiation + G100 10μg/Tumor | Part 2: Local Radiation + G100 10μg/Tumor+Pembrolizumab 200mg | Part 2: Local Radiation, G100 20 μg/Tumor in Large Tumors | Part 3: Local Radiation + G100 20μg/Tumor | Part 4: G100 20μg/Tumor and Pembrolizumab 200mg
Number analyzed (Participants) | 3 | 3 | 13 | 13 | 4 | 14 | 1
Participants | 0 | 0 | 0 | 2 | 0 | 1 | 0

3. Secondary Outcome: Overall Response Rate (ORR) by Immune-related Response Criteria (irRC)
Description: Overall response rate was defined as the number and percent of participants with best overall response of immune-related complete response (irCR) or immune-related partial response (irPR). irRC requires confirmatory restaging to determine if tumor size increase is due to true progression instead of immune inflammation and that new tumors add to tumor size calculations are not determinants of progressive disease by themselves. An immune-related Complete Response (irCR) is the disappearance of all tumors, measured or unmeasured, and no new tumors; an immune-related Partial Response (irPR) is a ≥50% drop in tumour burden from baseline as defined by the irRC; and immune-related Progressive Disease (irPD) is a ≥25% increase in tumour burden from the lowest level recorded. Everything else is considered immune-related Stable Disease (irSD). Tumor staging using bi-dimensional measurements was performed by CT or MRI.
Time Frame: Up to approximately 42 months
Population: The analysis population included all enrolled participants without major protocol deviations, who received at least 1 injection of G100, and had baseline and at least 1 post-baseline disease assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Local Radiation + G100 5μg/Tumor | Part 1: Local Radiation + G100 10μg/Tumor | Part 2: Local Radiation + G100 10μg/Tumor | Part 2: Local Radiation + G100 10μg/Tumor+Pembrolizumab 200mg | Part 2: Local Radiation, G100 20 μg/Tumor in Large Tumors | Part 3: Local Radiation + G100 20μg/Tumor | Part 4: G100 20μg/Tumor and Pembrolizumab 200mg
Number analyzed (Participants) | 3 | 3 | 13 | 13 | 4 | 14 | 1
Participants
  Complete Response (irCR) | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Partial Response (irPR) | 1 | 2 | 3 | 6 | 1 | 6 | 0
  Stable Disease (irSD) | 2 | 1 | 8 | 6 | 3 | 7 | 1
  Progressive Disease (irPD) | 0 | 0 | 2 | 1 | 0 | 1 | 0

4. Secondary Outcome: Clinical Benefit Rate (CBR) Using Immune-related Response Criteria (irRC)
Description: Clinical benefit rate (CBR) was defined as the number and percent of participants with best overall response of complete response, partial response or stable disease (irCR+irPR+irSD). Clinical response was assessed by Immune-related Response Criteria (irRC) using bi-dimensional measurements as a preliminary indication of efficacy. irRC requires confirmatory restaging to determine if tumor size increase is due to true progression instead of immune inflammation and that new tumors add to tumor size calculations are not determinants of progressive disease by themselves. An immune-related Complete Response (irCR) is the disappearance of all tumors, and no new tumors; an immune-related Partial Response (irPR) is a ≥50% drop in tumor burden from baseline; and immune-related Progressive Disease (irPD) is a ≥25% increase in tumor burden from the lowest level recorded. Everything else is considered immune-related Stable Disease (irSD). Tumor staging by CT or MRI was performed.
Time Frame: Up to approximately 42 months
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percent of participants
Arm/Group | Part 1: Local Radiation + G100 5μg/Tumor | Part 1: Local Radiation + G100 10μg/Tumor | Part 2: Local Radiation + G100 10μg/Tumor | Part 2: Local Radiation + G100 10μg/Tumor+Pembrolizumab 200mg | Part 2: Local Radiation, G100 20 μg/Tumor in Large Tumors | Part 3: Local Radiation + G100 20μg/Tumor | Part 4: G100 20μg/Tumor and Pembrolizumab 200mg
Number analyzed (Participants) | 3 | 3 | 13 | 13 | 4 | 14 | 1
Percent of participants | 100 [29.2 to 100] | 100 [29.2 to 100] | 84.6 [54.6 to 98.1] | 92.3 [64.0 to 99.8] | 100 [39.8 to 100] | 92.9 [66.1 to 99.8] | 100 [2.5 to 100]

5. Secondary Outcome: Clinical Benefit Rate (CBR) Using International Working Group (IWG) Criteria
Description: Clinical benefit rate (CBR) will be defined as the number and percent of participants with best overall response of complete response, partial response or stable disease (CR+PR+SD). The IWG criteria (Cheson et al 2014) for a CR is a complete radiologic response (target nodes/nodal masses must regress to ≤1.5 cm in longest transverse diameter (LDi), no extralymphatic sites of disease, and no new tumors. A PR is a ≥50% decrease in SPD (sum of the product of the perpendicular diameters for multiple tumors) of up to 6 target measurable nodes and extranodal sites, spleen must have regressed by >50% in length beyond normal, and no new tumors. Stable disease is a <50% decrease from baseline in SPD of up to 6 dominant, measurable nodes and extranodal sites; no criteria for progressive disease are met, and no new tumors.
Time Frame: Up to approximately 42 months
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Part 1: Local Radiation + G100 5μg/Tumor | Part 1: Local Radiation + G100 10μg/Tumor | Part 2: Local Radiation + G100 10μg/Tumor | Part 2: Local Radiation + G100 10μg/Tumor+Pembrolizumab 200mg | Part 2: Local Radiation, G100 20 μg/Tumor in Large Tumors | Part 3: Local Radiation + G100 20μg/Tumor | Part 4: G100 20μg/Tumor and Pembrolizumab 200mg
Number analyzed (Participants) | 3 | 3 | 13 | 13 | 4 | 14 | 1
Percentage of participants | 100 [29.2 to 100] | 100 [29.2 to 100] | 84.6 [54.6 to 98.1] | 92.3 [64.0 to 99.8] | 100 [39.8 to 100] | 78.6 [49.2 to 95.3] | 100 [2.5 to 100]

6. Secondary Outcome: Duration of Response (DOR) by Immune-related Response Criteria (irRC)
Description: Duration of response (DOR) was defined as the time interval between the date of the earliest qualifying confirmed/unconfirmed response using irRC and the date of disease progression (PD) or death for any cause, whichever occurs first. DOR in months was calculated as: (date of PD or death minus date of first confirmed/unconfirmed irCR/CR or irPR/PR + 1)/30.4375. DOR analysis included only participants with confirmed/unconfirmed response of irCR/irPR using irRC. Immune-related Progressive Disease (irPD) is a ≥25% increase in tumor burden from the lowest level recorded. Summary of DOR including median was estimated using the Kaplan-Meier method in each treatment group.
Time Frame: Up to approximately 42 months
Population: The analysis population included all enrolled participants who received at least 1 injection of G100 after standard local radiation and had a confirmed/unconfirmed response of irCR/irPR using irRC.
Measure: Median (Full Range); unit: Months
Arm/Group | Part 1: Local Radiation + G100 5μg/Tumor | Part 1: Local Radiation + G100 10μg/Tumor | Part 2: Local Radiation + G100 10μg/Tumor | Part 2: Local Radiation + G100 10μg/Tumor+Pembrolizumab 200mg | Part 2: Local Radiation, G100 20 μg/Tumor in Large Tumors | Part 3: Local Radiation + G100 20μg/Tumor | Part 4: G100 20μg/Tumor and Pembrolizumab 200mg
Number analyzed (Participants) | 1 | 1 | 3 | 4 | 1 | 5 | 0
Months | 1.8 [1.8 to 1.8] | 15.6 [15.6 to 15.6] | NA [NA to NA] — NA = Median DOR and DOR upper and lower limits were not reached as there was no progressive disease by the time of last disease assessment. | 18.4 [3.8 to 27.2] | NA [NA to NA] — NA = Median DOR and DOR upper and lower limits were not reached as there was no progressive disease by the time of last disease assessment. | 5.6 [2.8 to 16.1] |

7. Secondary Outcome: Duration of Clinical Benefit by Immune-related Response Criteria (irRC)
Description: Duration of clinical benefit was defined as the time interval between the date of the earliest qualifying confirmed/unconfirmed best response using irRC and the date of progression disease (PD) or death for any cause, whichever occurred first. Duration of clinical benefit in months was calculated as: (date of PD or death - date of first confirmed/unconfirmed irCR/irPR or irSD + 1)/30.4375. Duration of clinical benefit included only participants with confirmed/unconfirmed response of irCR/irPR or irSD using irRC. For participants who were alive without documentation of disease progression following the qualifying response, duration of clinical benefit was censored following the same rule defined for PFS. Summary of duration of clinical benefit including median was estimated using the Kaplan Meier method in each treatment group.
Time Frame: Up to approximately 42 months
Population: The analysis population included all enrolled participants who received at least 1 injection of G100 after standard local radiation and had a confirmed/unconfirmed response of irCR/irPR or irSD using irRC.
Measure: Median (Full Range); unit: Months
Arm/Group | Part 1: Local Radiation + G100 5μg/Tumor | Part 1: Local Radiation + G100 10μg/Tumor | Part 2: Local Radiation + G100 10μg/Tumor | Part 2: Local Radiation + G100 10μg/Tumor+Pembrolizumab 200mg | Part 2: Local Radiation, G100 20 μg/Tumor in Large Tumors | Part 3: Local Radiation + G100 20μg/Tumor | Part 4: G100 20μg/Tumor and Pembrolizumab 200mg
Number analyzed (Participants) | 3 | 3 | 11 | 12 | 4 | 13 | 0
Months | 2.5 [1.8 to 3.4] | 20.8 [0.0 to 26.0] | 6.9 [0.0 to 16.2] | 9.2 [2.8 to 27.2] | 7.2 [0.0 to 20.1] | 4.3 [0.0 to 20.0] |

8. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS was defined as time from date of first study treatment to date of first disease progression by irRC criteria, symptomatic deterioration, or death due to any cause, whichever occurs first. Progression-free survival in months is calculated as: (date of first progression, symptomatic deterioration, or death (any reason) - date of first dose +1)/30.4375. The irRC modification required a PD confirmation no less than 4 weeks from first documentation of PD; once confirmed, the date of progression was defined as date of the first PD. Participants without progression, symptomatic deterioration, or death were censored at the date of the last tumor assessment. Immune-related Progressive Disease (irPD) is a ≥25% increase in tumor burden from the lowest level recorded. Summary of PFS including median was estimated using the Kaplan-Meier method in each treatment group.
Time Frame: Up to approximately 42 months
Population: as for outcome 3
Measure: Median (Full Range); unit: Months
Arm/Group | Part 1: Local Radiation + G100 5μg/Tumor | Part 1: Local Radiation + G100 10μg/Tumor | Part 2: Local Radiation + G100 10μg/Tumor | Part 2: Local Radiation + G100 10μg/Tumor+Pembrolizumab 200mg | Part 2: Local Radiation, G100 20 μg/Tumor in Large Tumors | Part 3: Local Radiation + G100 20μg/Tumor | Part 4: G100 20μg/Tumor and Pembrolizumab 200mg
Number analyzed (Participants) | 3 | 3 | 13 | 13 | 4 | 14 | 1
Months | 4.9 [3.7 to 5.3] | 22.6 [1.9 to 27.7] | 7.4 [1.7 to 33.7] | 11.1 [1.9 to 32.5] | 9.8 [1.9 to 21.9] | 7.7 [1.4 to 22.6] | NA [NA to NA] — NA = Median PFS and PFS upper and lower limits were not reached as there was no disease progression or death by time of last disease assessment.

9. Secondary Outcome: Overall Survival (OS)
Description: Overall Survival (OS) was defined as the time from date of first study treatment to death due to any cause. Overall survival in months was calculated as: (date of death - date of first dose) +1)/30.4375. Participants who were alive at the end of study were censored at the last date the participant was known to be alive or data analysis cutoff date, whichever was earlier. Summary of OS including median was estimated using the Kaplan-Meier method in each treatment group.
Time Frame: Up to approximately 42 months
Population: as for outcome 3
Measure: Median (Full Range); unit: Months
Arm/Group | Part 1: Local Radiation + G100 5μg/Tumor | Part 1: Local Radiation + G100 10μg/Tumor | Part 2: Local Radiation + G100 10μg/Tumor | Part 2: Local Radiation + G100 10μg/Tumor+Pembrolizumab 200mg | Part 2: Local Radiation, G100 20 μg/Tumor in Large Tumors | Part 3: Local Radiation + G100 20μg/Tumor | Part 4: G100 20μg/Tumor and Pembrolizumab 200mg
Number analyzed (Participants) | 3 | 3 | 13 | 13 | 4 | 14 | 1
Months | NA [NA to NA] — NA = Median OS and OS upper and lower limits were not reached as there was an insufficient number of deaths by time of last disease assessment. | NA [NA to NA] — NA = Median OS and OS upper and lower limits were not reached as there was an insufficient number of deaths by time of last disease assessment. | NA [NA to NA] — NA = Median OS and OS upper and lower limits were not reached as there was an insufficient number of deaths by time of last disease assessment. | NA [NA to NA] — NA = Median OS and OS upper and lower limits were not reached as there was an insufficient number of deaths by time of last disease assessment. | NA [NA to NA] — NA = Median OS and OS upper and lower limits were not reached as there was an insufficient number of deaths by time of last disease assessment. | NA [NA to NA] — NA = Median OS and OS upper and lower limits were not reached as there was an insufficient number of deaths by time of last disease assessment. | NA [NA to NA] — NA = Median OS and OS upper and lower limits were not reached as there was an insufficient number of deaths by time of last disease assessment.

10. Secondary Outcome: Overall Tumor Response Based on irRC Abscopal Sites
Description: Abscopal tumor responses were assessed in non-treated, distal tumor sites. Clinical response was assessed by Immune-related Response Criteria (irRC) using bi-dimensional measurements as a preliminary indication of efficacy. irRC requires confirmatory restaging to determine if tumor size increase is due to true progression instead of immune inflammation and that new tumors add to tumor size calculations are not determinants of progressive disease by themselves. An immune-related Complete Response (irCR) is the disappearance of all tumors, measured or unmeasured, and no new tumors; an immune-related Partial Response (irPR) is a ≥50% drop in tumour burden from baseline as defined by the irRC; and immune-related Progressive Disease (irPD) is a ≥25% increase in tumour burden from the lowest level recorded. Everything else was considered immune-related Stable Disease (irSD). Tumor staging by CT or MRI was performed.
Time Frame: Up to approximately 42 months
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Local Radiation + G100 5μg/Tumor | Part 1: Local Radiation + G100 10μg/Tumor | Part 2: Local Radiation + G100 10μg/Tumor | Part 2: Local Radiation + G100 10μg/Tumor+Pembrolizumab 200mg | Part 2: Local Radiation, G100 20 μg/Tumor in Large Tumors | Part 3: Local Radiation + G100 20μg/Tumor | Part 4: G100 20μg/Tumor and Pembrolizumab 200mg
Number analyzed (Participants) | 3 | 3 | 13 | 13 | 4 | 14 | 1
Participants
  Complete Response (irCR) | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Partial Response (irPR) | 0 | 1 | 4 | 3 | 0 | 3 | 0
  Stable Disease (irSD) | 1 | 2 | 4 | 8 | 3 | 9 | 1
  Progressive Disease (irPD) | 1 | 0 | 4 | 2 | 1 | 2 | 0

11. Secondary Outcome: Time to Response for Complete Response and Partial Response Participants
Description: Time to Response for CR and PR participants was defined as time from date of first study treatment to the date of CR or PR response first documented. Complete Response (irCR) is the disappearance of all tumors, and no new tumors; an immune-related Partial Response (irPR) is a ≥50% drop in tumor burden from baseline. Time to response in months was calculated as: (date of first CR or PR minus date of first dose +1)/30.4375. Summary of Time to Response including median was estimated using Kaplan-Meier method in each treatment group.
Time Frame: Up to approximately 42 months
Population: The analysis population included all enrolled participants without major protocol deviations, who received at least 1 injection of G100, had baseline and at least 1 post-baseline disease assessment, and had a best response of CR or PR.
Measure: Median (Full Range); unit: Months
Arm/Group | Part 1: Local Radiation + G100 5μg/Tumor | Part 1: Local Radiation + G100 10μg/Tumor | Part 2: Local Radiation + G100 10μg/Tumor | Part 2: Local Radiation + G100 10μg/Tumor+Pembrolizumab 200mg | Part 2: Local Radiation, G100 20 μg/Tumor in Large Tumors | Part 3: Local Radiation + G100 20μg/Tumor | Part 4: G100 20μg/Tumor and Pembrolizumab 200mg
Number analyzed (Participants) | 1 | 2 | 3 | 6 | 1 | 6 | 0
Months | 1.9 [1.9 to 1.9] | 1.9 [1.9 to 1.9] | 2.3 [1.7 to 18.1] | 4.1 [2.2 to 14.1] | 2.6 [2.6 to 2.6] | 5.2 [1.9 to 7.3] |

12. Secondary Outcome: Time to Next Treatment (TTNT)
Description: Time to next treatment was defined as the time from the date of first study treatment to the start date of subsequent therapy after PD. Immune-related Progressive Disease (irPD) is a ≥25% increase in tumor burden from the lowest level recorded. Participants who did not receive subsequent therapy after PD were censored at the date of last contact or death. Summary of TTNT including median was estimated using the Kaplan-Meier method in each treatment group.
Time Frame: Up to approximately 42 months
Population: The analysis population included all enrolled participants without major protocol deviations, who received at least 1 injection of G100, had baseline and at least 1 post-baseline disease assessment, and had subsequent therapy with PD.
Measure: Median (Full Range); unit: Months
Arm/Group | Part 1: Local Radiation + G100 5μg/Tumor | Part 1: Local Radiation + G100 10μg/Tumor | Part 2: Local Radiation + G100 10μg/Tumor | Part 2: Local Radiation + G100 10μg/Tumor+Pembrolizumab 200mg | Part 2: Local Radiation, G100 20 μg/Tumor in Large Tumors | Part 3: Local Radiation + G100 20μg/Tumor | Part 4: G100 20μg/Tumor and Pembrolizumab 200mg
Number analyzed (Participants) | 3 | 1 | 8 | 6 | 1 | 6 | 0
Months | 5.4 [4.1 to 6.6] | NA [NA to NA] — NA = Median TTNT and TTNT upper and lower limits were not reached as there was an insufficient number of treatments by time of last assessment. | 12.7 [1.9 to 33.7] | NA [NA to NA] — NA = Median TTNT and TTNT upper and lower limits were not reached as there was an insufficient number of treatments by time of last assessment. | NA [NA to NA] — NA = Median TTNT and TTNT upper and lower limits were not reached as there was an insufficient number of treatments by time of last assessment. | NA [NA to NA] — NA = Median TTNT and TTNT upper and lower limits were not reached as there was an insufficient number of treatments by time of last assessment. |

ADVERSE EVENTS:
Time Frame: Up to approximately 42 months
Description: The analysis population included all enrolled and treated participants. Per protocol, disease progression of cancer under study was not considered an adverse event (AE) unless considered treatment-related. Medical Dictionary for Regulatory Activities (MedDRA) preferred terms "Neoplasm progression", "Malignant neoplasm progression" and "Disease progression" not related to study treatment were excluded as AEs. Part 5, G100 plus Rituximab, Dose Escalation: no participant was enrolled or dosed.
Arm/Group | Part 1: Local Radiation + G100 5μg/Tumor | Part 1: Local Radiation + G100 10μg/Tumor | Part 2: Local Radiation + G100 10μg/Tumor | Part 2: Local Radiation + G100 10μg/Tumor+Pembrolizumab 200mg | Part 2: Local Radiation, G100 20 μg/Tumor in Large Tumors | Part 3: Local Radiation + G100 20μg/Tumor | Part 4: G100 20μg/Tumor and Pembrolizumab 200mg
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 1/13 | 1/14 | 0/4 | 1/14 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 1/13 | 4/13 | 0/4 | 0/14 | 0/1
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 13/13 | 13/13 | 4/4 | 14/14 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: Local Radiation + G100 5μg/Tumor (N=3) | Part 1: Local Radiation + G100 10μg/Tumor (N=3) | Part 2: Local Radiation + G100 10μg/Tumor (N=13) | Part 2: Local Radiation + G100 10μg/Tumor+Pembrolizumab 200mg (N=13) | Part 2: Local Radiation, G100 20 μg/Tumor in Large Tumors (N=4) | Part 3: Local Radiation + G100 20μg/Tumor (N=14) | Part 4: G100 20μg/Tumor and Pembrolizumab 200mg (N=1)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Multiple fractures (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: Local Radiation + G100 5μg/Tumor (N=3) | Part 1: Local Radiation + G100 10μg/Tumor (N=3) | Part 2: Local Radiation + G100 10μg/Tumor (N=13) | Part 2: Local Radiation + G100 10μg/Tumor+Pembrolizumab 200mg (N=13) | Part 2: Local Radiation, G100 20 μg/Tumor in Large Tumors (N=4) | Part 3: Local Radiation + G100 20μg/Tumor (N=14) | Part 4: G100 20μg/Tumor and Pembrolizumab 200mg (N=1)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (2) | 2 (3) | 1 (4) | 0 (0) | 0 (0)
Blood loss anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymph node pain (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocardial fibrosis (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Ear congestion (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Diplopia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eyelid ptosis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Periorbital oedema (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (2) | 2 (4) | 2 (3) | 2 (2) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (2) | 1 (1) | 0 (0)
Dental caries (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 4 (4) | 0 (0) | 2 (2) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoaesthesia oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 6 (7) | 1 (2) | 3 (4) | 0 (0)
Rectal tenesmus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Administration site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (7) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Fatigue (General disorders) | 1 (1) | 2 (2) | 0 (0) | 4 (4) | 2 (2) | 3 (3) | 1 (1)
Feeling hot (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 1 (2) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Infusion site swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site bruising (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injection site discomfort (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site erythema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Injection site pain (General disorders) | 0 (0) | 0 (0) | 3 (5) | 1 (1) | 0 (0) | 2 (3) | 0 (0)
Injection site reaction (General disorders) | 0 (0) | 1 (1) | 1 (5) | 2 (4) | 0 (0) | 1 (8) | 0 (0)
Injection site swelling (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (4) | 2 (2) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Candida infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Helicobacter duodenitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes virus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Oesophagitis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rhinovirus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (5) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Expired product administered (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Radiation associated pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Radiation skin injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 3 (5) | 1 (1) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Blast cell count increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 1 (2) | 2 (5) | 1 (2) | 0 (0) | 0 (0)
Blood bilirubin decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (5) | 0 (0)
Blood creatinine decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Blood glucose increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Breath sounds abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemoglobin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 1 (1) | 3 (6) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 1 (1) | 2 (4) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (3) | 3 (5) | 0 (0) | 1 (2) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (7) | 2 (2) | 0 (0)
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypernatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 2 (3) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 2 (2) | 0 (0) | 0 (0)
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Carpal tunnel syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (3) | 0 (0) | 2 (3) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nystagmus (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Libido decreased (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Restlessness (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sleep disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary hesitation (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Epididymal cyst (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oedema genital (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Testicular atrophy (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Testis discomfort (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal inflammation (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 4 (5) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (4) | 0 (0) | 1 (1) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (3) | 3 (5) | 0 (0) | 0 (0) | 0 (0)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin swelling (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin texture abnormal (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diastolic hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Embolism (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (2) | 2 (4) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Systolic hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Varicose vein (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The study was terminated (halted prematurely) for business reasons.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor will have 30 days for review/ comment on any manuscripts from results of this clinical trial, and can request an additional 30 days in order to protect the Sponsor's confidential, proprietary data, and intellectual property rights. Abstracts, press releases, and other media presentations must also be forwarded to the Sponsor prior to release. No publication, manuscript, or other form of public disclosure shall contain any of the Sponsor's confidential/ proprietary information.

DOCUMENTS (2):
  • Study Protocol (2018-11-15): https://cdn.clinicaltrials.gov/large-docs/73/NCT02501473/Prot_000.pdf
  • Statistical Analysis Plan (2019-07-17): https://cdn.clinicaltrials.gov/large-docs/73/NCT02501473/SAP_001.pdf